CLINICAL TRIAL: NCT02134574
Title: Prospective Cohort Study of Clinical and Laboratory Data of Patients With Hemopathy in Languedoc-Roussillon
Brief Title: Prospective Cohort With Hemopathy in Languedoc-Roussillon
Acronym: HemoDiag
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9011
Record Dates: First submitted 2014-04-22; First posted 2014-05-09 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Hematologic Malignancy
Keywords: Lymphoma,; leukemia,; multiple myeloma,; hodgkin disease
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Leukemia; Multiple Myeloma; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hematologic malignancy: hematologic malignancy with a sampling of blood
  Interventions: Biological: hematologic malignancy

INTERVENTIONS:
Biological: hematologic malignancy — hematologic malignancy with a sampling of blood
  Other Names: hematologic malignancy with a sampling of blood

SUMMARY:
Prospective Cohort Study of clinical and laboratory data of patients with hemopathy.

DETAILED DESCRIPTION:
Prospective Cohort Study of clinical and laboratory data of patients with hemopathy in LR.

ELIGIBILITY:
Inclusion criteria:

* Age over 18
* Consultant or hospitalized patient for suspected malignant hemopathy and justifying further exploration or patient with a diagnosis of malignant hemopathy less than 6 months old at the time of signing the consent
* Having signed an informed consent
* Affiliated with a social security scheme

Exclusion criteria:

* Minor or major protected
* Patients who have received treatment for hematological pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient for suspected haematological disease and justifying further exploration
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-02; Primary Completion 2033-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Survival with 2 years | 2 years
  Prospective Cohort Study of clinical and biological data Analysis Biological, clinical and questionnaire EORTC_QLQ-C30

SECONDARY OUTCOMES:
Survival with 5 years | 5 years
  Prospective Cohort Study of clinical and biological data Analysis Biological, clinical and questionnaire EORTC_QLQ-C30
Survival with 10 years | 10 years
  Prospective Cohort Study of clinical and biological data Analysis Biological, clinical and questionnaire EORTC_QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: GUILLAUME CARTRON, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hematology department - UHMontpellier Saint éloi, Montpellier, France